CLINICAL TRIAL: NCT05918991
Title: Interventions for English Language Learners At-Risk for ADHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: Florida State University (Other); Nova Southeastern University (Other); University of South Florida (Other)
Responsible Party: Principal Investigator, Dr. Nicki Schatz, Research Associate Professor, Florida International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R324A210221
Record Dates: First submitted 2023-02-22; First posted 2023-06-26 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: English Language Learners; Classroom Behavioral Intervention; Language Intervention
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Motion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Individuals completing classroom behavioral observations are masked to participant intervention assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Language Intervention (Experimental): The language intervention will include 18 weeks of 20-25 minutes of intervention approximately 4 days per week. The language intervention is delivered via shared book reading and focuses on English language vocabulary development as well as development of syntax knowledge and expressive language.
  Interventions: Other: Language Intervention
- Daily Report Card (Experimental): The Daily Report Card group will receive the Daily Report Card intervention for 18 weeks.
  Interventions: Behavioral: Daily Report Card
- Combined Language and Daily Report Card (Experimental): Participants in this arm will receive a combination of the language intervention and the behavioral intervention. The interventions will be implemented simultaneously for 18 weeks.
  Interventions: Behavioral: Daily Report Card; Other: Language Intervention
- School As Usual (No Intervention): Participants in the School as Usual Arm will receive neither the Behavioral Intervention nor the Language Intervention. There will be no restrictions, however, on interventions or supports that students may receive outside of the study either implemented through standard school protocol or accessed by parents. Thus, the School as Usual Arm provides a real-world practice comparison for the three active treatment groups.

INTERVENTIONS:
Behavioral: Daily Report Card — Behavioral consultants will meet with teachers to review daily report card implementation and effective classroom management. The consultant collaborates with the teacher to identify specific behavioral goal targets for the student's DRC based on a review of teacher ratings and teacher description of key problem behaviors. After establishing the initial DRC, the consultant will review procedures with the teacher for scoring the DRC and, importantly, providing the student with effective and consistent performance feedback. The consultant will also make a plan with the teacher to review DRC progress and revise the DRC as needed. Consultants will also meet with parents to develop a plan for reinforcing the DRC at home. The DRC will be implemented for 18 weeks. The behavioral consultants will be available to teachers and parents throughout the duration of the intervention to assist with implementation and adjustment of target behaviors and goals.
  Arms: Combined Language and Daily Report Card; Daily Report Card
Other: Language Intervention — The intervention protocol to be provided in each grade level will include 18 weeks of 20-25 minutes of small-group intervention 4 days per week, for a total of 72 lessons. The fifth day per week will be allocated to make-up lessons for students absent earlier in the week to maximize opportunity for each participant to receive the full dosage of lessons. Half of these lessons in each grade will be allocated to Language in Motion implementation and the other half to Dialogic Reading. Dialogic Reading is designed to increase vocabulary knowledge through shared reading of picture books. The content involves reading of 9 children's books with 108 targeted vocabulary words. Language in Motion is designed to increase syntax and grammar knowledge using science manipulatives. Daily lessons are highly scripted to introduce primary syntax targets through narrative text. Manipulation props are used to reinforce syntax targets and basic science topics.
  Other Names: Dialogic Reading, Language in Motion
  Arms: Combined Language and Daily Report Card; Language Intervention

SUMMARY:
The goal of this clinical trial is to compare the effect of language and behavioral interventions for students who are English language learners and who have symptoms of attention-deficit/hyperactivity disorder (ADHD). The main question it aims to answer is:

- Which intervention is better for the students: the behavioral intervention, the language intervention, or a combination of the behavioral and language interventions?

Participants will be asked to do the following:

* Participants' parents and teachers will be asked to complete questionnaires about their behavior.
* Participants will be asked to complete tests assessing language, cognitive, and academic abilities.
* Members of the research team will complete classroom observations for the participating students.
* Participants will be randomly assigned to one of four groups: a school as usual group, a language group, a daily report card group, and a combined daily report card and language group.

  * If assigned to the language group, participants will receive an 18-week language intervention.
  * If assigned to the daily report card group, a behavioral consultant will work with participants' parents and teachers to set up a home-school behavior plan called a daily report card.
  * If assigned to the combined daily report card and language group, participants will receive both the language intervention and the daily report card.
  * If assigned to the school as usual group, participants will no study interventions.

Researchers will compare the language group, the daily report card group, the combined language and daily report card group, and the school as usual group to see which group has the best language learning and classroom behavior at the end of the program.

ELIGIBILITY:
Inclusion Criteria:

* Identified as an English Language Learner Level 1 through 4 by their school district
* Enrolled in kindergarten or 1st grade during the year of participation
* 6 or more symptoms of attention-deficit/hyperactivity disorder endorsed by parent or teacher
* Has a teacher who is willing to participate
* Has a parent or primary caregiver who is willing to participate

Exclusion Criteria:

* Participant has an active Individualized Education Plan for language or behavior
* Participant IQ is less than 70
* Participant is diagnosed with psychosis
* Participant is diagnosed with autism spectrum disorder with severity level 2 or greater or another pervasive developmental disorder
* Participant is enrolled in home-school

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Expressive One-Word Picture Vocabulary Test 4th Edition (EOWPVT-4) Score | Post-treatment (i.e., after completion of the 18-week treatment phase)
  The EOWPVT-4 (Martin & Brownell, 2011) consists of 190 items used to assess children's ability to verbally label illustrations of objects, actions, or concepts. Basal, based on child age, and ceiling (i.e., six consecutive incorrect responses) rules are used. Internal consistency (alpha) for ages 3-10 years ranges from .95 to .97, and split-half reliability, corrected for full length of the test, ranges from .96 to .98.
Word Classes 1 Subtest Score | Post-treatment (i.e., after completion of the 18-week treatment phase)
  Clinical Evaluation of Language Fundamentals-4th Edition (CELF-4), Word Classes 1 Subtest. The Word Classes I subtest of the CELF-4 includes 21 (ages 5 to 7 years) items used to assess children's ability to recognize and identify words that share a semantic relationship. The examiner says three or four words (e.g., porcupine, quills, ball) and the child correctly responds by saying how two of the words are related (i.e., Porcupines have quills.). All children begin at the first item, and a ceiling is established after seven consecutive incorrect responses. Internal consistency (alpha) for ages 5-11 years ranges from.85 to .92.
Sentence Structure Subtest Score | Post-treatment (i.e., after completion of the 18-week treatment phase)
  Clinical Evaluation of Language Fundamentals-4th Edition (CELF-4), Sentence Structure subtest. The CELF-4 Sentence Structure subtest consists of 26 items designed to assess the children's ability to comprehend spoken sentences of increasing length and syntactic complexity. Children listen to a sentence spoken by the examiner and select one picture out of four that illustrates the referential meaning of the sentence. All children begin at the first item and a ceiling is established after five consecutive incorrect responses. Internal consistency (alpha) for ages 5:0 - 8:11 years of age ranges from .64 to .76, and test-retest reliability for ages 6 - 7:11 years ranges from .67 to .74.
Syntax Construction Subtest Score | Post-treatment (i.e., after completion of the 18-week treatment phase)
  Comprehensive Assessment of Spoken Language (CASL), Syntax Construction subtest. The Syntax Structure subtest of the CASL consists of 56 items used to assess the children's ability to formulate and express sentences using a variety of morphosyntactic rules. While showing the child a picture in the stimulus manual, the examiner either reads one to three sentences with a phrase missing from the final sentence (e.g., "This is a small fish. This is a ___." [big fish]) or gives the child a directive to say something related to the picture (e.g., "The man found the hat. Where was it?" [on the table]). Basal, based on child age, and ceiling (i.e., five consecutive incorrect responses) rules are used. Internal consistency (alpha) for ages 5-10 years ranges from .82 to .90, and test-retest reliability for ages 5-7 years is .79 and for ages 8-11 years is .74.
Concepts and Following Directions Subtest Score | Post-treatment (i.e., after completion of the 18-week treatment phase)
  Clinical Evaluation of Language Fundamentals-4th Edition (CELF-4), Concepts and Following Directions subtest. The Concepts and Following Directions subtest of the CELF-4 consists of 54 items used to assess children's abilities to interpret and follow directions of increasing length and complexity (e.g., names, characteristics, and order of mention) using logical operations (e.g., before/after, tallest, etc.). Basal, based on child age, and ceiling (i.e., seven consecutive incorrect responses) rules are used. Internal consistency (alpha) ranges from .73 to .92, and test-retest reliability ranges from .67 to .88.
Oral Comprehension Subtest Score | Post-treatment (i.e., after completion of the 18-week treatment phase)
  Woodcock-Johnson Tests of Achievement, 3rd Edition (WJ-III), Oral Comprehension subtest. The Oral Comprehension subtest of the WJ-III consists of 34 items that assess children's ability to comprehend short, audio-recorded or orally presented passages to complete an oral close task. The child hears a sentence followed by two beeps (for audio-recorded presentation) at which time the child provides a single word to finish the sentence. Basal, based on child grade, and ceiling (i.e., six consecutive items are responded to incorrectly) rules are used. Median internal consistency for children ages 5-19 years is .80, and one-year, test-retest reliability for children 4-7 years of age is .82.
Frequency counts of off-task behavior | Post-treatment (i.e., after completion of the 18-week treatment phase)
  This outcome measure is collected via systematic direct observations of student classroom behavior by trained observers masked to treatment condition. The score is a frequency count of off-task behaviors during 30-minute observation periods. Because this is a count variable, the minimum value is zero and there is no maximum value. Higher scores indicate worse outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Florida International University, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
The final data file will include (a) raw item-level data (where applicable to recreate analyses) with appropriate variable and value labels (b) all computed variables created during setup and scoring, and (c) all scale scores for the demographic, behavioral, and assessment or any other data used in a final analytic model.